CLINICAL TRIAL: NCT07031440
Title: Digital Delivery of Living Well With COPD for Patient Education and Self-management - a Mixed-method Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Cantonal Hospital of St. Gallen (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STD0007385
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- digital LWWCOPD (Other)
  Interventions: Behavioral: digital LWWCOPD

INTERVENTIONS:
Behavioral: digital LWWCOPD — LWWCOPD (Living well with COPD) contains six modules conventionally delivered by trained LWWCOPD Coaches. For the digital delivery the six modules are as closely adapted to the conventional LWWCOPD program as possible to make the two approaches comparable. Participants can access the digital LWWCOPD application by a weblink using a smartphone, tablet or desktop computer. Since the program duration of the conventional LWWCOPD is 6 weeks (one module per week), patients will be instructed to complete the digital LWWCOPD also within 6 weeks at their own pace, although completion within 12 weeks (3 months) is still possible. Modules can be repeated as chosen by the user. In contrast to the conventional delivery, the online delivery of LWWCOPD does not preview face-to-face contact between participants and healthcare providers, however if needed additional phone calls or meetings are still possible.

SUMMARY:
COPD (Chronic Obstructive Pulmonary Disease) is a common lung disease. People suffering from COPD typically experience shortness of breath, coughing, and mucus production. The condition is usually treated with medication, but it is equally important that patients are well-informed about COPD and receive guidance on how to live with it.

The currently available program, "Living well with COPD (LWWCOPD)," is a patient education and self-management program offered on-site in healthcare institutions (such as the Lung League) over six sessions across six weeks. Studies have shown that participating in this program can improve quality of life and overall health, and COPD patients who have completed it tend to require hospitalization less frequently.

However, not all patients who could benefit from the program are able to attend in person-either due to the fixed schedule or because traveling to the training site is too difficult. Therefore, this study aims to determine whether the digital version of the "Living well with COPD" program is equally effective and perhaps more convenient for some patients. The digital version closely mirrors the existing program and consists of various modules that provide information about COPD and practical strategies for managing the disease in daily life. Only once its effectiveness is scientifically proven can the digital version be implemented in Switzerland for COPD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Diagnosis of COPD (any stage and severity)
3. Able to speak/read/understand German or French
4. Access to a cell phone, tablet or personal desktop computer with active internet access
5. Willing and able to understand and provide written informed consent
6. Current or recent enrolment in a pulmonary rehabilitation program is permitted

Exclusion Criteria:

1. Inability to follow the procedures/instructions of the study or to participate in the intervention (e.g. due to language or cognitive barriers, psychological disorders, physical reasons)
2. Patients already having completed the conventional LWWCOPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in HRQoL (Health-Related Quality of Life) | From enrollment to the end of intervention at 3 months
  Change in HRQoL, assessed by the Chronic Respiratory Disease Questionnaire (CRQ) from baseline (before start with digital LWWCOPD program) to three months follow-up (after completion of digital LWWCOPD program)